CLINICAL TRIAL: NCT00574223
Title: Double-Blind, Placebo-Controlled Study to Investigate Safety, Tolerability, Immunogenicity and Clinical Efficacy of a Specific Immunotherapy Combining Allergen With CYT003-QbG10 (CYT005-AllQbG10) in Adult Patients With Perennial Allergic Rhinoconjunctivitis Due to House Dust Mite Allergy
Brief Title: A Study to Investigate an Immunomodulatory Therapy in Adult Patients With Perennial Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Philipp Mueller, MD, Head of Clinical Development, EVP, Cytos Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT005-AllQbG10 04
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Perennial Allergic Rhinoconjunctivitis; House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy | interventions — CYT003-QbG10; Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: CYT005-AllQbG10 (combination of house dust mite allergen extract with CYT003-QbG10)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: House dust mite allergen extract in combination with CYT003-QbG10-placebo

INTERVENTIONS:
Drug: CYT005-AllQbG10 (combination of house dust mite allergen extract with CYT003-QbG10) — subcutaneous injections at 8 visits
  Arms: Arm 1
Drug: House dust mite allergen extract in combination with CYT003-QbG10-placebo — subcutaneous injections at 8 visits
  Arms: Arm 2

SUMMARY:
The purpose of the study is to test the efficacy of the combination treatment AllQbG10 in patients with perennial allergic rhinoconjunctivitis due to house dust mite allergy in a double-blind placebo-controlled setting

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate perennial allergic rhinoconjunctivits due to hypersensitization towards house dust mite allergens

Exclusion Criteria:

* Clinically relevant other allergies (perennial or seasonal) that could potentially interfere with the patient's study treatment schedule or assessments
* Use of any concomitant medication that could affect the patient's study treatment response or assessment results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Conjunctival provocation test with allergen and rhinoconjunctivitis symptoms in daily life | about 1.5 hours on 4 occasions over 1 year

SECONDARY OUTCOMES:
Safety and tolerability of the study treatment by collection of adverse events | about 30 min. at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Mueller, MD, Study Director — Cytos Biotechnology
Locations (1):
- Cytos Biotechnology (Sponsor's Headquarter), Schlieren, Switzerland